CLINICAL TRIAL: NCT01565746
Title: Uncontrolled, Open-label, Non-randomized Phase I Study to Investigate Safety, Biodistribution, Radiation Dosimetry and Pharmacokinetics of a Single Dose of BAY88-8223 in Japanese Patients With Castration-resistant Prostate Cancer and Bone Metastases
Brief Title: Safety, Biodistribution, Radiation Dosimetry and Pharmacokinetics Study of BAY88-8223 in Japanese Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15354
Record Dates: First submitted 2012-03-01; First posted 2012-03-29 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Prostatic Neoplasms
Keywords: BAY88-8223; radium-223 dichloride; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Radium-223 dichloride [50 kBq/kg] (Experimental)
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)
- Radium-223 dichloride [100 kBq/kg] (Experimental)
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)
- Radium-223 dichloride [expansion] (Experimental)
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Radium-223 dichloride (Xofigo, BAY88-8223) 50 kBq/kg
  Arms: Radium-223 dichloride [50 kBq/kg]
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Radium-223 dichloride (Xofigo, BAY88-8223) 100 kBq/kg
  Arms: Radium-223 dichloride [100 kBq/kg]
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Expansion arm: Radium-223 dichloride (Xofigo, BAY88-8223) 50 kBq/kg
  Arms: Radium-223 dichloride [expansion]

SUMMARY:
This is an uncontrolled, open-label, non-randomized Phase I study to investigate safety, biodistribution, radiation dosimetry and pharmacokinetics of a single dose of BAY88-8223 in Japanese patients with castration-resistant prostate cancer and bone metastases.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 20 years of age
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Presents with at least 2 bone metastases, confirmed by scintigraphic imaging within the previous 4 weeks
* Patients who has failed initial hormonal therapy using either an orchiectomy or a Gonadotropin releasing hormone (GnRH) agonist in combination with an antiandrogen must first progress through antiandrogen withdrawal prior to being eligible. The minimum timeframe to document failure of anti-androgen withdrawal will be four weeks
* Progressive castration resistant metastatic disease
* Castrate level of testosterone (<50 ng/dL), treatment to maintain castrate levels of testosterone must be continued

Exclusion Criteria:

* Has received an investigational drug in the 4 weeks before or is scheduled to receiving one during or in the 8 weeks after study drug administration.
* Has received chemo-, immuno-, or radiotherapy within the last 4 weeks prior to entry in the study, or has not recovered from acute adverse events as a result of such therapy
* Has received prior hemibody external radiotherapy
* Has a need for immediate external radiotherapy
* Has received systemic radiotherapy with radium-223, strontium-89, samarium-153, rhenium-186 or rhenium-188 for the treatment of bony metastases within the last 24 weeks prior to administration of study drug
* When receiving bisphosphonates, has changed the dose within 4 weeks before administration of study drug

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with Critical toxicities | Up to day 28
  Critical toxicities (using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0) will be defined as the occurrence of one or more of the following drug-related toxicities: 1) ≥Grade 3 non-hematologic toxicity, 2) Grade 3 neutropenia with fever, 3) Grade 4 neutropenia that failed to recover to grade 2 or less after treatment with Granulocyte colony-stimulating factor (GCSF) within 2 weeks, 4) Grade 4 thrombocytopenia
Maximum drug concentration in blood after single dose administration (Cmax) of BAY88-8223 for blood samples | up to 72 hours
Area under the concentration - time curve (AUC) of BAY88-8223 for blood samples | up to 72 hours

SECONDARY OUTCOMES:
Changes in prostate specific antigen (PSA) | baseline, up to 12 weeks
Overall Survival | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Japan (3):
  - Kashiwa, Chiba
  - Yokohama, Kanagawa
  - Sayama, Osaka

REFERENCES:
- [Result] Yoshida K, Kaneta T, Takano S, Sugiura M, Kawano T, Hino A, Yamamoto T, Shizukuishi K, Kaneko M, Zurth C, Inoue T. Pharmacokinetics of single dose radium-223 dichloride (BAY 88-8223) in Japanese patients with castration-resistant prostate cancer and bone metastases. Ann Nucl Med. 2016 Aug;30(7):453-60. doi: 10.1007/s12149-016-1093-8. Epub 2016 Jun 7. PMID 27272279
- [Derived] Uemura H, Uemura H, Matsubara N, Kinuya S, Hosono M, Yajima Y, Doi T. Safety and efficacy of radium-223 dichloride in Japanese patients with castration-resistant prostate cancer and bone metastases. Int J Clin Oncol. 2017 Oct;22(5):954-963. doi: 10.1007/s10147-017-1130-1. Epub 2017 May 6. PMID 28478485